CLINICAL TRIAL: NCT05786209
Title: A Single-Center, Four Week Usage Clinical Study to Evaluate the Tolerance and Efficacy of a Whole-Body Balm on Newborn Babies
Brief Title: A Study of a Whole-Body Balm on Newborn Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCSSKB005124; CCSSKB005124 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Therapeutic Irrigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole-body Balm + Wash and Shampoo (Experimental): Parent participant will be instructed to apply the whole-body balm on the newborn baby's whole body (excluding the mouth, eyes, diaper area, and scalp) two times per day (morning and evening), and to cleanse the newborn baby with the wash and shampoo at least once per week and no more than three times per week up to Day 28.
  Interventions: Other: Whole-body Balm; Other: Wash and Shampoo

INTERVENTIONS:
Other: Whole-body Balm — Balm will be applied to cover newborn's entire body (while avoiding the mouth, eyes, diaper area, and scalp), and gently massaged onto the skin until the balm is fully absorbed.
Other: Wash and Shampoo — Wash and shampoo will be used to cleanse newborn baby using an "in tub" bathing method.

SUMMARY:
The purpose of this study is to evaluate the skin tolerance, instrumental efficacy, and perceived product efficacy of a whole-body balm on newborns (0-28 days old).

ELIGIBILITY:
Inclusion Criteria:

Newborn participants only:

* Male or Female
* 0 to 3 months old, targeting at least 15 subjects in the 0 - 28 days age range at time of enrollment.
* Has Parent Participant-reported Natural Skin tone/skin Color As Follows, including: (a) Skin tones "Pale/fair to light white" and/or "White to light beige" approximately 10 participants; (b) Skin tones "Beige to light tan/light olive" and/or "Medium tan/medium olive to light brown" approximately 10 participants; (c) Skin tones "Medium brown to dark brown" and/or "Darkest brown to darkest black" approximately 10 participants
* Full term (37 plus weeks of gestation, both vaginal and Caesarean mode of delivery can be included) newborn

Newborn participant and parent participant:

* Generally, in good health based on medical history reported by the parent participant

Parent participant only:

* Able to read, write, speak, and understand English
* At least 18 years old and is the parent (adoptive or biological), legal guardian, and primary caregiver of the newborn participant
* Has signed the informed consent document (ICD) including Health Insurance Portability and Accountability Act (HIPAA) disclosure
* Intends to complete the study and is willing and able to follow all study instructions

Exclusion Criteria:

Newborn participant only:

* Presents with a skin condition that may influence the outcome of the study or increase risk to the newborn participant (example , psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema, or active skin cancer)
* Has a family history of (defined as having a biological parent or full sibling with) eczema/atopic dermatitis
* Has been bathed within 3 hours prior to Visit 1
* Has a clinical grade greater than 0 for rash/irritation, or greater than or equal to 1 for any of the other clinically assessed tolerance parameters at Visit 1

Newborn participant and parent participant:

* Has known allergies or adverse reactions to common topical skincare products
* Has self-reported (for the parent participant) or parent participant reported (for the newborn participant) Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication
* Is taking a medication that would mask an AE or confound the study results, including (a) Immunosuppressive or steroidal drugs within 3 months before Visit 1; (b) Non-steroidal anti-inflammatory drugs within 5 days before Visit 1; (C) Antihistamines within 2 weeks (14 days) before Visit 1

Ages: 0 Days to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Change From Baseline After 4 Weeks of Product Use in Clinical and Parental Evaluations of Skin tolerance Measures | Change from baseline after 4 weeks
  Change from baseline after 4 weeks of product use in clinical and parental evaluations of skin tolerance measures will be reported. The clinical and parental evaluations of tolerance will be recorded on paper source documentation.

SECONDARY OUTCOMES:
Change From Baseline After 7 Days of Product Use in Clinical and Parental Evaluations of Skin Tolerance Measures | Change from baseline after 7 days
  Change from baseline after 7 days of product use in clinical and parental evaluations of skin tolerance measures will be reported. The clinical and parental evaluations of tolerance will be recorded on paper source documentation.
Change From Baseline After 7 Days of Product Use in Corneometer and Transepidermal Water Loss (TEWL) Measurements | Change from baseline after 7 days
  Change from baseline after 7 days of product use in Corneometer and TEWL measurements will be reported. The Corneometer measures moisture content in the stratum corneum by an electrical capacitance method. Readings are proportional to the dielectric constant of the surface layers of the skin, and the results are displayed in arbitrary "Corneometer units" ranging from 0 to 120, with increasing values corresponding to more hydrated skin. TEWL is a equipment with open chamber TEWL probes to measure the TEWL of the skin. The non-invasive probe contains two sensors that measure the temperature and relative humidity at two fixed points along the axis normal to the skin surface.
Change From Baseline After 4 Weeks of Product Use in Corneometer and Transepidermal Water Loss (TEWL) Measurements | Change from baseline after 4 weeks
  Change from baseline after 4 weeks of product use in Corneometer and TEWL measurements will be reported. The Corneometer measures moisture content in the stratum corneum by an electrical capacitance method. Readings are proportional to the dielectric constant of the surface layers of the skin, and the results are displayed in arbitrary "Corneometer units" ranging from 0 to 120, with increasing values corresponding to more hydrated skin. TEWL is a equipment with open chamber TEWL probes to measure the TEWL of the skin. The non-invasive probe contains two sensors that measure the temperature and relative humidity at two fixed points along the axis normal to the skin surface.
Number of Response Options for Each Question in the Parental Questionnaire | Day 28
  Number of response options for each question in the parental questionnaire will be reported. Parental questionnaire will be completed by the parent participants which include the questions about "how much do you agree after using balm" where 1 indicates 'strongly disagree', 2 indicates 'somewhat disagree', 3 indicates ;neither agree or disagree', 4 indicates 'somewhat agree', 5 indicates 'strongly agree'.
Percentage of All Response Options for Each Question in the Parental Questionnaire | Day 28
  Percentage of all response options for each question in the parental questionnaire will be reported. parental questionnaire will be completed by the parent participants which include the questions about "how much do you agree after using balm" where 1 indicates 'strongly disagree', 2 indicates 'somewhat disagree', 3 indicates ;neither agree or disagree', 4 indicates 'somewhat agree', 5 indicates 'strongly agree'.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, M.D., Principal Investigator — Cenexel JBR
Locations (1):
- CenExcel JBR, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] https://www.courage-khazaka.de/en/scientific-products/all-products/16-wissenschaftliche-produkte/alle-produkte/183-corneometer-e.
- See also: Redacted CSR Synopsis with Disclaimer — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSSKB005124&attachmentIdentifier=30ec3d13-90e5-4e19-820a-0f351ee1d334&fileName=CCSSKB005124_CSR_Synopsis_English.pdf&versionIdentifier=